CLINICAL TRIAL: NCT04863924
Title: Accelerating Lung Cancer Diagnosis Through Liquid Biopsy
Acronym: ACCELERATE
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Lung Health Foundation (Unknown); The Princess Margaret Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20-5915
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced NSCLC: Patients with radiologic evidence of advanced (unresectable stage III or IV) non-small cell lung cancer
  Interventions: Diagnostic Test: Liquid Biopsy

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy — All patients will have a liquid biopsy with ctDNA molecular profiling

SUMMARY:
This study will assess the utility of liquid biopsy to accelerate the time to treatment for patients with newly diagnosed advanced non-small cell lung cancer, compared to the conventional diagnostic pathway of molecular testing of tumour tissue after imaging and biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Lung RAMP Multidisciplinary Cancer Conference or study team confirms radiologic (clinical) evidence of advanced, unresectable lung cancer;
2. Measurable disease (presumed malignant) by RECIST 1.1;
3. Age ≥18 years;
4. Ability to provide written informed consent;
5. Diagnostic biopsy and molecular profiling ordered or planned. Patients remain eligible even if biopsy or tumour testing later fails or is deemed not feasible.

Exclusion Criteria:

1. Pregnancy;
2. Concurrent active malignancy except for localized non-melanomatous skin cancer or non-invasive cervical cancer. Any previous cancer (excluding NSCLC) must have been treated more than 2 years prior to study entry with no current evidence of active disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the UHN Lung Cancer Rapid Assessment & Management Program (Lung RAMP) with radiologic evidence of advanced (unresectable stage III or IV) non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to treatment | Up to 18 Months
  The time to treatment decision (TLB) in the study cohort by liquid (TL) and tissue biopsy (TB) is measured from the date of referral to the earliest date of receiving a liquid or tissue biopsy report indicating actionable genomic aberrations, or TLB = min (TL, TB). The time to treatment decision using tissue biopsy alone (TB) will be collected in a chart-review comparison cohort (patients referred in the previous 12 months that meet the eligibility criteria). The time to treatment decision by liquid biopsy (TLB) vs by tissue biopsy alone (TB) will be compared.

SECONDARY OUTCOMES:
Time to treatment - non-smoker subgroup | Up to 18 Months
  Measure the time to treatment, using the same parameters as the primary outcome measure, in a subgroup of patients with advanced non-squamous NSCLC with a smoking history of ≤15 pack years.
Turnaround time | Up to 18 Months
  Calculate the time (in days) from the date of request for testing to the report date for both liquid biopsy and tissue biopsy.
Concordance between liquid and tissue | Up to 18 Months
  Count the number of actionable targets identified by liquid biopsy and by tissue biopsy, by patient, that were in agreement.
Costs of upfront use of liquid biopsy vs standard tissue profiling | Up to 24 Months
  A cost-effectiveness model will be developed comparing the initial use of liquid biopsy versus the current standard of tissue biopsy and profiling.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Canada

REFERENCES:
- [Derived] Garcia-Pardo M, Czarnecka-Kujawa K, Law JH, Salvarrey AM, Fernandes R, Fan ZJ, Waddell TK, Yasufuku K, Liu G, Donahoe LL, Pierre A, Le LW, Gunasegaran T, Ghumman N, Shepherd FA, Bradbury PA, Sacher AG, Schmid S, Corke L, Feng J, Stockley T, Pal P, Rogalla P, Pipinikas C, Howarth K, Ambasager B, Mezquita L, Tsao MS, Leighl NB. Association of Circulating Tumor DNA Testing Before Tissue Diagnosis With Time to Treatment Among Patients With Suspected Advanced Lung Cancer: The ACCELERATE Nonrandomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2325332. doi: 10.1001/jamanetworkopen.2023.25332. PMID 37490292